CLINICAL TRIAL: NCT04981483
Title: Long-term Follow-up of the Cases Who Underwent Conservative Surgery for Placenta Previa Accreta
Brief Title: Conservative Surgery for Placenta Accreta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mohammed mahmoud samy, assisstant professor of obstetrics and gynaecology, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11784
Record Dates: First submitted 2021-07-06; First posted 2021-07-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Any age and parity with placenta accreta spectrum (Experimental): After removal of the placenta, grasping the cervix from the both lips and one from each side of the cervical canal at the level of the internal os, each uterine angle and grasped the remaining lower uterine segment and Nelaton catheter was inserted inside the cervical canal to avoid closing the cervix with sutures of the uterine incision.Closing the uterine incision;taking suture at the lateral angle of the cervix and suturing it to the lower edge of the uterine angle, then another continuous suture was attached to the upper edge of the uterine incision angle[outside in-in out then out in-in out] and the same technique was repeated on the other side (cervico-isthmic sutures). controlling bleeding from the inner surface of the remaining lower uterine segment was done by 2-3 interrupted sutures between the lower uterine segment and the anterior cervical lip. closing of the uterine incision in continuous non-locking manner
  Interventions: Procedure: conservative surgery for uterus in placenta accreta

INTERVENTIONS:
Procedure: conservative surgery for uterus in placenta accreta — After removal of the placenta, grasping the cervix from the both lips and one from each side of the cervical canal at the level of the internal os, each uterine angle and grasped the remaining lower uterine segment and Nelaton catheter was inserted inside the cervical canal to avoid closing the cervix with sutures of the uterine incision.Closing the uterine incision;taking suture at the lateral angle of the cervix and suturing it to the lower edge of the uterine angle, then another continuous suture was attached to the upper edge of the uterine incision angle[outside in-in out then out in-in out] and the same technique was repeated on the other side (cervico-isthmic sutures). controlling bleeding from the inner surface of the remaining lower uterine segment was done by 2-3 interrupted sutures between the lower uterine segment and the anterior cervical lip. closing of the uterine incision in continuous non-locking manner

SUMMARY:
A stepwise surgical approach for conservative management of placenta previa accreta.

DETAILED DESCRIPTION:
a stepwise surgical approach for conservative management of placenta previa accreta to preserve women's uterus and to evaluate the efficacy and safety of this approach in controlling postpartum hemorrhage including intrapartum hemorrhage associated with conservative management.

ELIGIBILITY:
Inclusion Criteria:

* Any age.
* Any parity.
* Previous one or more cesarean delivery.
* Placenta previa accreta diagnosis confirmed by gray scale & color flow Doppler ultrasound in 3rd trimester. All participants had undergone abdominal ultrasound showing placenta previa anterior completely covering the internal os, with criteria suggestive of invasion by U/S

Exclusion Criteria:

* women with medical disorder
* women with bleeding tendency

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
incidence rate of conserving woman's uterus | intraoperative
  success rate of conservative surgery for placenta accreta

SECONDARY OUTCOMES:
number of units of packed red blood cells , Fresh Frozen Plasma transfused ,postoperative haemoglobin | till 48 hours postpartum
  to assess blood loss
incidence rate of cesarean hysterectomy needed | intraoperative and 48 hours postpartum
  failure of conservation , increase in blood loss
incidence of puerperal sepsis | till 6 weeks postpartum
  temperature chart every 6 hours in 1st 48 hours postpartum then follow up visits 2 weeks and 6 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud ghaleb, lecturer, Study Director — ainshams university faculty of medicine
Locations (1):
- Ain SHams Maternity Hospital, Cairo, Abbaseya, Egypt

IPD SHARING:
Plan to Share IPD: No